CLINICAL TRIAL: NCT03836105
Title: Cemiplimab Survivorship Epidemiology (CASE) Study
Brief Title: CemiplimAb Survivorship Epidemiology
Acronym: CASE
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R2810-ONC-1806
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Basal Cell Carcinoma
Keywords: Locally Advanced CSCC (laCSCC); Metastatic CSCC (mCSCC); Locally Advanced BCC (laBCC); Metastatic BCC (mBCC)
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — cemiplimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: This group will enroll patients with advanced (defined as locally advanced or metastatic [nodal or distant]) CSCC.
  Interventions: Drug: cemiplimab
- Group 2: This group will enroll patients with advanced (defined as locally advanced or metastatic [nodal or distant]) BCC.
  Interventions: Drug: cemiplimab

INTERVENTIONS:
Drug: cemiplimab — No investigational agents will be provided to enrolled patients by the sponsor as part of this study. Patients will have recently initiated or be planning to initiate treatment with commercially available cemiplimab for advanced CSCC or advanced BCC in a real-world setting according to respective label indications. In addition to cemiplimab, patients may receive other therapies as deemed necessary by their physicians for the treatment of CSCC or BCC or comorbid conditions.
  Other Names: REGN2810; Libtayo

SUMMARY:
The objectives of the study are:

* To describe the effectiveness of cemiplimab 350 mg administered every 3 weeks (Q3W) for treatment of patients with advanced (defined as locally advanced or metastatic [nodal or distant]) cutaneous squamous cell carcinoma (CSCC) and patients with advanced (defined as locally advanced or metastatic [nodal or distant]) basal cell carcinoma (BCC) in real-world clinical settings
* To evaluate the safety of cemiplimab based on incidence of treatment related immune-related adverse events (irAEs), infusion related reactions (IRRs), and treatment related serious adverse reactions (TSARs) in patients with advanced CSCC and patients with advanced BCC receiving cemiplimab treatment in real world clinical settings
* To describe patient experience, including patient reported quality of life (QOL) and functional status, and clinician reported performance status in a real-world setting for patients with advanced CSCC and patients with advanced BCC
* To describe baseline characteristics that could potentially be associated with health-related outcomes for patients with advanced CSCC and patients with advanced BCC undergoing treatment with cemiplimab
* To describe patients who receive cemiplimab as treatment for CSCC or BCC in a real-world setting
* To describe real-world use patterns of cemiplimab for CSCC and BCC
* To investigate the long-term effects and effectiveness of cemiplimab in patients with advanced CSCC or advanced BCC
* To describe the effectiveness of cemiplimab in immunosuppressed and immunocompetent patients with advanced CSCC or advanced BCC, regardless of etiology, per available data
* To describe the effectiveness of cemiplimab after prior exposure to radiation therapy for CSCC per available data
* To describe the effectiveness of cemiplimab as a first-line (1L) or later systemic treatment in patients with advanced CSCC, regardless of etiology, per available data
* To describe the effectiveness of cemiplimab in patients with advanced BCC based on treatment patterns (reason for discontinuation, treatment exposure, etc) of prior Hedgehog inhibitor (HHI) usage

ELIGIBILITY:
Key Inclusion Criteria:

* Eligible for treatment with and prescribed cemiplimab for advanced CSCC or advanced BCC in accordance with approved prescribing information as described in the protocol

Key Exclusion Criteria:

* Receiving cemiplimab for an indication other than advanced CSCC or advanced BCC
* Any condition that, in the opinion of the investigator, may interfere with patient's ability to participate in the study
* Patients concurrently participating in any study including administration of any investigational drug (including cemiplimab) or procedure (including survival follow up)

Note: Other protocol defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in this study will include men and women ≥18 years of age who have recently initiated, or who plan to initiate treatment with commercially available cemiplimab for laCSCC/mCSCC or laBCC/mBCC in a real-world setting.
Sampling Method: Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 36 months
  The rate of complete responses (CR) or partial responses (PR), as assessed by investigators
Disease control rate (DCR) | Up to 36 months
  Percentage of patients who have achieved CR, PR or stable disease (SD) to cemiplimab as assessed by investigators
Duration of response (DOR) | Up to 36 months
  Time from the time of initial response until documented tumor progress, death, or initiation of non-cemiplimab CSCC or BCC treatment
Time to response | Up to 36 months
  Time from date of first admission of cemiplimab to the initial response
Progression free survival (PFS) | Up to 36 months
  Time from the date of first administration of cemiplimab to progression or death from any cause, whichever occurs first
Overall Survival (OS) | Up to 36 months
  Time from the date of first administration of cemiplimab to the date of death due to any cause
Time to treatment failure (TTTF) | Up to 36 months
  Time from date of first administration of cemiplimab to treatment discontinuation for disease progression, treatment toxicity, or death
Disease specific death (DSD) | Up to 36 months
  Rate of death cause by or related to underlying CSCC or BCC as assessed by investigators
Number of patients with metastatic vs locally advanced cancer summarized every three weeks | Up to 36 months
  Pattern of recurrence
Immune related adverse events (irAEs) | Up to 36 months
  Per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5
Infusion related reactions (IRRs) | Up to 36 months
  NCI-CTCAE v5
Treatment related serious adverse reactions (SARs) | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceutical, Inc.
Locations (52):
- United States (50):
  - Oncology Specialties, PC - Clearview Cancer Institute, Huntsville, Alabama
  - Dignity Health St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - CARTI Cancer Center, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - Harbor-UCLA/LA Biomedical Research Institute, Los Angeles, California
  - St. Mary's Medical Center, San Francisco, California
  - Regeneron Research Facility, Stanford, California
  - University of Colorado, Aurora, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Regional Cancer Care Associates, LLC, Manchester, Connecticut
  - Integrity Clinical Research, Delray Beach, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Regeneron Research Facility, Largo, Florida
  - Regeneron Research Facility, Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Lewis Hall Singletary Oncology Center at John D. Archbold Memorial Hospital, Thomasville, Georgia
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Reid Oncology Association, Richmond, Indiana
  - CHRISTUS Highland Cancer Treatment Center, Shreveport, Louisiana
  - Baltimore Veterans Affairs Medical Center, Baltimore, Maryland
  - Frederick Health, Frederick, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Southeast Nebraska Hematology & Oncology Consultants, PC, Lincoln, Nebraska
  - Optum Cancer Care, Las Vegas, Nevada
  - Regeneron Research Facility, Elizabeth, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Regeneron Research Facility, New York, New York
  - Regeneron Research Facility, Nyack, New York
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - Montefiore Hospital, The Bronx, New York
  - Oncology Specialists of Charlotte, PA, Charlotte, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Texas Oncology-Amarillo Cancer Center, Amarillo, Texas
  - Texas Oncology, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
- Puerto Rico (2):
  - Pan-American Center for Oncology Trials, LLC, Rio Piedras
  - FDI Clinical Research, San Juan

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Park SJ, Ellison DM, Weight R, Homsi J, Rabinowits G, Ruiz ES, Strasswimmer J, Simmons J, Panella T, Quek RG, Pouliot JF, Khushalani NI. CASE (CemiplimAb-rwlc Survivorship and Epidemiology): a study in advanced basal cell carcinoma. Future Oncol. 2025 Feb;21(4):431-436. doi: 10.1080/14796694.2024.2448416. Epub 2025 Jan 11. PMID 39797702
- [Derived] Migden MR, Chandra S, Rabinowits G, Chen CI, Desai J, Seluzhytsky A, Sasane M, Campanelli B, Chen Z, Freeman ML, Ibrahim SF, Khushalani NI, Andria M, Ruiz E. CASE (CemiplimAb-rwlc Survivorship and Epidemiology) study in advanced cutaneous squamous cell carcinoma. Future Oncol. 2020 Feb;16(4):11-19. doi: 10.2217/fon-2019-0762. Epub 2020 Jan 17. PMID 31951149